CLINICAL TRIAL: NCT05477771
Title: The Correlation Between the Cross-sectional Area of the Long Head of the Biceps Tendon and the Tear Position in Patients With Rotator Cuff Tears
Brief Title: The Cross-sectional Area of the Long Head of the Biceps Tendon and the Rotator Cuff Tear Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0028
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Tears
Keywords: long head of the bicep tendon; rotator cuff tear; cross-sectional area
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anterior tear group (Experimental): The rotator cuff was divided into three parts according to the arthroscopic discovery: (1) the anterior part which contained the subsacpularis and one third of the suprascapularis forward; (2) the middle part which contained the two thirds of the suprascapularis backward and one third of the subscapularis forward; (3) the posterior part which contained two thirds of subscapularis backward and teres minor. The patients with rotator cuff tear at the anterior part were categorized in the anterior tear group.
  Interventions: Procedure: Arthroscopic rotator cuff repair
- Middle tear group (Experimental): The rotator cuff was divided into three parts according to the arthroscopic discovery: (1) the anterior part which contained the subsacpularis and one third of the suprascapularis forward; (2) the middle part which contained the two thirds of the suprascapularis backward and one third of the subscapularis forward; (3) the posterior part which contained two thirds of subscapularis backward and teres minor. The patients with rotator cuff tear at the middle part were categorized in the middle tear group.
  Interventions: Procedure: Arthroscopic rotator cuff repair
- Posterior tear group (Experimental): The rotator cuff was divided into three parts according to the arthroscopic discovery: (1) the anterior part which contained the subsacpularis and one third of the suprascapularis forward; (2) the middle part which contained the two thirds of the suprascapularis backward and one third of the subscapularis forward; (3) the posterior part which contained two thirds of subscapularis backward and teres minor. The patients with rotator cuff tear at the posterior part were categorized in the posterior tear group.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — The rotator cuff tears were repaired under arthroscopy. A subacromial decompression was performed in all patients. Then the long head of the biceps with severe lesions were treated by tenotomy while the others were reserved according to the surgeon's judgment during the surgery.

SUMMARY:
The main aim and scope of this study is making measurement and comparison of the cross-sectional area of the long head of the biceps tendon(LHBT) in the patients suffered form rotator cuff tear with different tear positions, and making observation and comparison of the impairment type of the LHBT in the patients suffered from rotator cuff tear with different tear positions. The results may identify the influence of the tear position on the LHBT.

ELIGIBILITY:
Inclusion Criteria:

* partial or full-thickness but reparable rotator cuff tear;
* small- to large-sized rotator cuff tears being defined by DeOrio and Cofied4;
* no improvements after at least 1 month of conservative treatment such as NSAIDs or corticosteroid injection.

Exclusion Criteria:

* massive rotator cuff tears being defined by DeOrio and Cofied;
* patients with osteoarthritis of the glenohumeral joint;
* trauma or a history of surgery at the shoulder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-07-29 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-22 (Estimated)

PRIMARY OUTCOMES:
Pre-operative measurement of the cross-sectional area of the long head of bicep tendon | Pre-operative
  According to the pre-operative MRI scan, two sites of the long head of biceps tendon were measured by the Image-Pro Plus 6.0 software. One was the plane that passed the center of the glenoid cavity, the other one was the plane that passed the distal border of the glenoid cavity. The contour of the long head of biceps tendon was traced and the area was calculated by the software according to the MRI's scale.

SECONDARY OUTCOMES:
Post-operative measurement of the cross-sectional area of the long head of bicep | 2 months after the surgery
  According to the MRI scan 2 months after the surgery, two sites of the long head of biceps tendon were measured by the Image-Pro Plus 6.0 software. One was the plane that passed the center of the glenoid cavity, the other one was the plane that passed the distal border of the glenoid cavity. The contour of the long head of biceps tendon was traced and the area was calculated by the software according to the MRI's scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No